CLINICAL TRIAL: NCT03423511
Title: CRYSTAL Study: A Multi-Center, Randomized, Controlled Trial to Demonstrate the Safety and Effectiveness of the MiStent II for the Revascularization of Coronary Arteries.
Brief Title: Trial to Demonstrate the Safety and Effectiveness of the MiStent II for the Revascularization of Coronary Arteries.
Acronym: CRYSTAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Micell Technologies (Industry)
Collaborators: Baim Institute for Clinical Research (Other); North American Science Associates Inc. (Unknown); Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIS-US-2017-01
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease
Keywords: MiStent; Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Disease; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: MiStent group vs. the Xience/Promus group.
Who Masked: Participant
Masking Description: This is a single-blind trial, such that the patient or patient's family will NOT be told which stent they have received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MiStent II Coronary Artery Stent (Experimental): Implantation of a coronary artery stent in an all-comers population, including patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions
  Interventions: Device: MiStent II coronary artery stent
- Xience or Promus Coronary Artery Stents (Active Comparator): Implantation of a coronary artery stent in an all-comers population, including patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions
  Interventions: Device: Xience or Promus coronary artery stents

INTERVENTIONS:
Device: MiStent II coronary artery stent — Implantation of a coronary stent patient with stable and unstable coronary artery disease including non-ST-Elevated Myocardial Infarction
  Arms: MiStent II Coronary Artery Stent
Device: Xience or Promus coronary artery stents — Implantation of a coronary stent patient with stable and unstable coronary artery disease including non-ST-Elevated Myocardial Infarction
  Arms: Xience or Promus Coronary Artery Stents

SUMMARY:
To compare MiStent to either the Xience or Promus stents.with the primary objective being to assess the safety and efficacy of the MiStent in a patient population requiring revascularization of de novo obstructive lesions of coronary arteries in patients with stable and unstable coronary artery disease (CAD) including non ST-Elevation Myocardial Infarction (NSTEMI)

DETAILED DESCRIPTION:
The CRYSTAL study is a prospective, multi-center, randomized (1:1), single-blinded and controlled, investigational device exemption trial to test the non-inferiority of MiStent to commercially available "everolimus" drug eluting stents (Xience and Promus stents).

Patients with coronary artery disease (CAD) that qualify for percutaneous coronary intervention (PCI) with stenting will be screened per the protocol inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age
2. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
3. Subject is eligible for percutaneous coronary intervention (PCI)
4. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia
5. Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
6. Subject is willing to comply with all protocol-required follow-up evaluation

   Angiographic Inclusion Criteria (visual estimate):
7. Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.50 mm and ≤3.50 mm
8. Target lesion(s) must be able to be treated with a single stent and the target lesion length must be ≤27 mm (by visual estimate).

   NOTE: Only lesion lengths that have both the control and comparable investigational stent lengths available at the same time are eligible for enrollment.
9. Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1 and one of the following:

   1. Stenosis ≥70% or;
   2. Abnormal fractional flow reserve (FFR) defined as <0.80 or;
   3. Abnormal stress or imaging stress test or;
   4. Elevated biomarkers prior to the procedure
10. Coronary anatomy is likely to allow delivery of a study device to the target lesions(s)
11. The first lesion treated must be successfully predilated/pretreated

Exclusion Criteria:

1. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation MI (STEMI)
2. Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
3. Subject has received an organ transplant or is on a waiting list for an organ transplant
4. Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
5. Planned PCI (including staged procedures) or CABG after the index procedure
6. Subject previously treated at any time with intravascular brachytherapy in the target vessel(s)
7. Subject has a known allergy to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g., Cobalt-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin)
8. Subject has one of the following (as assessed prior to the index procedure):

   1. Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months
   2. Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
   3. Planned procedure that may cause non-compliance with the protocol or confound data interpretation
9. Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin, or other anticoagulation therapy) for indications other than acute coronary syndrome
10. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
11. Subject has a white blood cell (WBC) count < 3,000 cells/mm3
12. Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
13. Subject is on dialysis or has baseline glomerular filtration rate (GFR) of <30 ml/min
14. Subject has a history of bleeding diathesis, active peptic ulcer or gastrointestinal (GI) bleed, or coagulopathy or will refuse blood transfusions
15. Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
16. Subject has severe symptomatic heart failure (i.e., Left Ventricular Ejection Fraction (LVEF) <30%))
17. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
18. Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
19. Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
20. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

    Angiographic Exclusion Criteria (visual estimate):
21. Planned treatment of a single lesion with more than 1 stent
22. Planned treatment of more than 3 lesions
23. Planned treatment of lesions in more than 2 major epicardial vessels
24. Planned treatment of more than 2 lesions in a single major epicardial vessel
25. Subject has 2 target lesions in the same vessel that are separated by less than 15 mm (by visual estimate)
26. Target lesion(s) is located in the left main or unprotected left
27. Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate
28. Target lesion(s) is located within a saphenous vein graft or an arterial graft
29. Target lesion(s) will be accessed via a saphenous vein graft or arterial graft
30. Target lesion(s) with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
31. Target lesion(s) treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
32. Target lesion(s) is restenotic from a previous stent implantation or study stent would overlap with a previous stent
33. Subject has been treated with any type of PCI (i.e., balloon angioplasty, stent, cutting balloon atherectomy) within 24 hours prior to the index procedure
34. Significant thrombus, present in the target vessel (by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | through 12-month visit
  Any occurrence of Target Lesion Failure (TLF)
  TLF is defined as:
  Cardiac death, or Target vessel myocardial infarction (TV-MI, Q-wave and non Q-wave), or Ischemia driven target lesion revascularization.

SECONDARY OUTCOMES:
Device success | Index Procedure
  Successful delivery and deployment of the study stent to the target vessel, without balloon rupture or stent embolization with post procedure diameter stenosis of < 30% (by visual estimation) in the Target Lesion.
Technical success | Index Procedure
  Achieving a final diameter stenosis of <30% (by visual estimation) in the target lesion using any combination of stents or devices allowed per protocol.
Procedural success | Index Procedure
  Post-procedure diameter stenosis <30% (by visual estimation) in all target lesions and the absence of in-hospital MI, TVR, or cardiac death.
Composite Endpoint POCE | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  POCE defined as all-cause death, any MI, or any revascularization
Composite Endpoint MACE | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  MACE defined as all-cause death, any MI, or any TVR
Composite Endpoint TVF | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  TVF defined as cardiac death, TV MI, or clinically indicated TVR
Composite Endpoint TLF | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  TLF defined as cardiac death, TV MI or Ischemia driven TLR
Mortality | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  Mortality including All death, Cardiac death, and Non-cardiac death (vascular and non-cardiovascular)
Myocardial Infarction | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  Myocardial Infarction including All MI, TV-MI, and Non-TV-MI
Revascularization | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  Revascularization including Target Lesion revascularization (TLR) (any, clinically- indicated TLR, non-clinically indicated TLR), Target Vessel revascularization (TVR) (any, clinically- indicated TVR, non-clinically indicated TVR), Non-TV revascularization, and Any revascularization
Stent thrombosis rates | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  Stent thrombosis rates according to ARC classification: ST - Early (Acute, Sub-acute), Late, Very Late; ST - Definite, Probable, Possible
Serious Adverse Events (SAEs) | prior to discharge, at 1-, 6- and 12-months and annually thereafter through 5 years' follow-up
  * All SAEs through 12 months' post-index procedure
  * All device related SAEs from 12 months through 5 years' post-index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mauri, MD, MSc, Study Chair — Brigham and Women's Hospial; Dean Kereiakes, MD, Principal Investigator — The Christ Hospital; David Kandzari, MD, Principal Investigator — Piedmont Heart Institute

IPD SHARING:
Plan to Share IPD: No